CLINICAL TRIAL: NCT01828853
Title: Maternal and Neonatal Outcomes After Membrane Sweeping
Acronym: Stripping
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Other Study IDs: Kabiri-Stripping-HMO-CTIL
Record Dates: First submitted 2013-01-30; First posted 2013-04-11 (Estimated); Last update posted 2013-04-11 (Estimated); Status verified 2013-03

CONDITIONS: Sepsis; Infection
Keywords: Membrane sweeping; Membrane stripping; Maternal outcomes; Neonatal outcomes
MeSH Terms: conditions — Sepsis; Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No

SUMMARY:
This study aim to estimate maternal and neonatal outcomes after membrane sweeping in different group of patients.

DETAILED DESCRIPTION:
Sweeping of the membranes is a simple technique usually performed during vaginal examination, in order to initiate labour by increasing local production of prostaglandins.

ELIGIBILITY:
Inclusion Criteria:

* Women with a singleton pregnancy and confirmed cephalic presentation at or after 37 weeks of gestation who are candidate for vaginal delivery were eligible for the study

Exclusion Criteria:

* Women with a multiple pregnancy, nonreassuring cardiotocogram, meconium stained amniotic fluid, major fetal anomalies, HELLP (hemolysis, elevated liver enzymes, and low platelets) syndrome, or severe preeclampsia and signs of intrauterine infections were not eligible.
* women who are not candidates for vaginal delivery: placenta previa, breech presentation, planned repeat cesarean.

Ages: 17 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: All women presenting to the Maternal-fetal unit who are 37+ weeks gestation
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2013-04; Primary Completion 2013-08 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Neonatal sepsis | Neonates will be followed for the duration of hospital stay, an expected average of 2-3 days

SECONDARY OUTCOMES:
Neonatal infection | Neonates will be followed for the duration of hospital stay, an expected average of 2-3 days
  Neonates with two or more of the following signs: Altered behaviour or responsiveness, Altered muscle tone (floppiness), Feeding difficulties, Feed intolerance (vomiting, excessive gastric aspirates, abdominal distension), Abnormal heart rate (bradycardia or tachycardia), Signs of respiratory distress, Hypoxia (central cyanosis or reduced oxygen saturation level), Jaundice, Apnoea, Signs of neonatal encephalopathy, Seizures, Need for cardio-pulmonary resuscitation, Low-temperature (lower than 36°C), High-temperature (higher than 38°C), Signs of shock, Unexplained excessive bleeding, thrombocytopenia or abnormal coagulation, Oliguria, Altered glucose homeostasis (hypoglycaemia or hyperglycaemia), Metabolic acidosis, Local signs of infection.

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel, Jerusalem, Israel